CLINICAL TRIAL: NCT04853563
Title: Comparison of High VErsus Low Positive End-Expiratory Pressure in Mechanically Ventilated Patients With Acute Heart Failure (HELP-AFH) : Open-label Randomized Controlled Multi-center Pilot Study
Brief Title: Comparison of PEEP in Acute Decompensated Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Seok Kim, professor of medicine, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC_2021_0433
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Heart Decompensation; Mechanical Ventilation Pressure High
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High PEEP (Experimental): Immediate after initiation of invasive mechanical ventilation and randomization, the PEEP level is set to be at 8 centimetre of water with an inspired oxygen fraction (FiO2) between 0.21 and 0.6. Thereafter, the PEEP level is adjusted to 1 centimetre of water higher to a minimum PEEP level of 10 with every 30 minutes.
  Interventions: Other: PEEP
- Low PEEP (Active Comparator): Immediate after initiation of invasive mechanical ventilation and randomization, the PEEP level is set to be at 5 centimetre of water with an inspired oxygen fraction (FiO2) between 0.21 and 0.6. In this arm, the PEEP level is adjusted to 1 centimetre of water lower to a minimum PEEP level of 3 with every 30 minutes while maintaining a partial pressure of arterial blood oxygen above 65 millimeter of mercury or oxygen saturation >92% with pulse oxymetry.
  Interventions: Other: PEEP

INTERVENTIONS:
Other: PEEP — High PEEP targeted to 10 cmH2O to be maintained during the period of mechanical ventilation compared with low PEEP maintaining 3-5 cmH2O

SUMMARY:
Little is known about optimal level of positive end-expiratory pressure (PEEP) in patiens who recieved invasive mechanical ventilation for acute decompensated heart failure. We therefore sought to compare clinical outcome according to low versus high PEEP.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who was diagnosed with congestive heart failure and objective evidence of pulmonary congestion (pulmonary edema on simple chest radiography or positive B-line on lung ultrasonography AND elevated B-type natriuretic peptide or N-terminal pro-brain natriuretic peptide level) as a reason for invasive mechanical ventilation
2. Age over 19 years old
3. Subject who agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the clinical site.

Exclusion Criteria:

1. Subject who are on mechanical circulatory support (ECMO, intra-aortic balloon pump, VAD) at the time of randomization
2. Subject who has cardiac abnormality that requires emergent or urgent percutaneous or surgical valvular procedure
3. Subject who are on vasoactive or inotropic agents at least moderate dose defined as vasoactive-inotropic score >10
4. Isolated preload-dependent cardiac dysfunction (isolated right ventricular failure, right ventricular infarction, constrictive pericarditis, cardiac tamponade, severe pulmonary hypertension without LV dysfunction)
5. Predominant right ventricular failure defined as following; clinical evidence of right ventricular failure by attending physician's discretion including hepatojugular reflux, Kussmaul sign, cardiac liver cirrhosis, hepato/splenomegaly, acites, thronmbocytopenia, etc.
6. Subject who are not on mechanical ventilation before open heart surgery
7. Subject who received unwitness cardiopulmonary rescucitation (CPR) or witness CPR lasting more than 30 minutes
8. Subject who was already diagnosed or is suspected to have hypertophic cardiomyopathy with significant left ventricular outflow tract (LVOT) obstruction
9. Subject with intracranial hemorrahge or ischemic stroke at the time of randomization
10. Subject with irreversible neurologic damage or irreversible hepatic failure
11. Invasive mechanical ventilation lasting more than 24 hours preceding endotracheal intubation
12. Subject with underlying chronic obstructive pulmonary disease (GOLD classification III or IV) or restrictive pulmonary disease (e.g. interstitial lung disease)
13. Subject with impaired consciousness that can not perform self coughing and need suction to maintain adequate airway patency
14. Pregnant and/or lactating women
15. Subject with life expectancy less than a year
16. Subject who is not suitable to enrollment by investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free day at 28-day | up to 28-day
  Starting at the day of randomization, and the days on non-invasive ventilation do not count. Successful extubation is defined as at least 24 hours wihtout reintubation independent of invasive assisted ventilation in survivor. Non-survivor within 28 days: ventilator-free day counted as 0, ventilator-free day among only survivor at 28-day will be counted for primary endpoint.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hyun J, Kim IC, Kim AR, Lee HJ, Lee SE, Yun SC, Kim MS. Comparison of High Versus Low Positive End-Expiratory Pressure in Mechanically Ventilated Patients With Acute Heart Failure: Rationale and Design of the HELP-AHF Trial. Int J Heart Fail. 2025 Apr 23;7(2):79-84. doi: 10.36628/ijhf.2025.0014. eCollection 2025 Apr. PMID 40519712